CLINICAL TRIAL: NCT06165978
Title: Physical Activity Coaching in Patients with Post-COVID-19. a Randomised Clinical Trial.
Brief Title: Physical Activity Coaching in Patients with Post-COVID-19
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: In response to recruitment difficulties, the study has been reclassified as a pilot phase. This adjustment will allow for an in-depth evaluation of feasibility and procedural refinements before considering a larger-scale trial.
Sponsor: University of Alcala (Other)
Collaborators: Colegio Profesional de Fisioterapeutas de la Comunidad de Madrid (Unknown)
Responsible Party: Principal Investigator, María José Yuste Sánchez, Associate Professor, Co-founder, and Co-Principal Investigator of the Physiotherapy in Women's Health Research Group - FPSM, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEID/2023/3/072
Record Dates: First submitted 2023-12-11; First posted 2023-12-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Post-COVID-19 Syndrome
Keywords: physical activity; physical activity coaching; post-COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Blood Glucose Self-Monitoring; Educational Status; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical activity coaching - Experimental group (Experimental): The experimental group intervention consists of a 12-week physical activity coaching program informed by the literature (CRD42021253066). The intervention is conducted at participants' home or within the community, delivered remotely (mostly) and face-to-face, and encompasses several behaviour change components (mandatory: self-monitoring, goal setting/review, education, feedback, contact; optional: exercise, reports, support meeting, group activities).
  Interventions: Behavioral: Self-monitoring; Behavioral: Goal setting and review; Behavioral: Education; Behavioral: Feedback; Behavioral: Contact; Behavioral: Exercise; Behavioral: Report; Behavioral: Social support; Behavioral: Group activities; Behavioral: World Health Organization recommendations for being physically active
- Usual care - Control group (Other): The control group intervention runs parallel to the experimental group for 12 weeks, conducted at participants' home or within the community, and consists of usual management (i.e., World Health Organization's recommendations for being physically active).
  Interventions: Behavioral: World Health Organization recommendations for being physically active

INTERVENTIONS:
Behavioral: Self-monitoring — pedometer/activity band provided to each participant
  Arms: Physical activity coaching - Experimental group
Behavioral: Goal setting and review — Goal setting and review (weekly: +15% of the previous week's average daily steps or walking time, or +1000 steps/day or +10 minutes walking - to be specified)
  Arms: Physical activity coaching - Experimental group
Behavioral: Education — Educational sessions (face-to-face: providing a manual/explanatory brochure of the intervention; remote: addressing symptom pathophysiology, symptom management, among other topics)
  Arms: Physical activity coaching - Experimental group
Behavioral: Feedback — Daily or weekly feedback for patients (emotional/social support)
  Arms: Physical activity coaching - Experimental group
Behavioral: Contact — Contact with patients (face-to-face: for assessments; on remote: 1 -messages: for therapists' daily/weekly feedback or patient reports; 2 - calls: to adjust weekly goals or address doubts or issues)
  Arms: Physical activity coaching - Experimental group
Behavioral: Exercise — Exercise based on patient preference, explaining how to identify moderate intensity (HRmax=64-76%, Borg 3-6) or vigorous intensity (HRmax=77-95%; Borg 7-8) and monitoring safety parameters (StO2>88%, HRmax<96%, Borg<9)
  Arms: Physical activity coaching - Experimental group
Behavioral: Report — Daily or weekly reporting for therapists (messages)
  Arms: Physical activity coaching - Experimental group
Behavioral: Social support — Support meetings (in-person), parallel to educational sessions
  Arms: Physical activity coaching - Experimental group
Behavioral: Group activities — Group activities (e.g., walking on familiar routes - parks, monumental areas, etc.)
  Arms: Physical activity coaching - Experimental group
Behavioral: World Health Organization recommendations for being physically active — World Health Organization's recommendations to maintain physical activity levels (i.e., 150-300 minutes/week of moderate to vigorous intensity physical activity; a weekly average of 10,000 steps/day or 100-120 minutes walking, which implies maintaining a pace of 100 steps/minute - corresponding to the average cadence across different age and gender groups).

SUMMARY:
This randomized clinical trial aims to compare the effects of a 12-week behavioral physical activity intervention (i.e., physical activity coaching) with usual care (i.e., World Health Organization recommendations for being physically active) in patients with post-COVID-19 (i.e., patients who suffered from COVID-19 at any degree of severity in acute phase and experience symptoms for at least three months after discharge).

This study aims to answer the following question:

1) Which are the effects of a physical activity coaching intervention compared with usual care in patients post-COVID-19 in the short-, middle- and long-term?

DETAILED DESCRIPTION:
Patients will be invited to participate via phone calls, and those interested will be scheduled to obtain their written informed consent and undergo a baseline assessment.

Afterwards, they will be randomized into an experimental group and a control group. In the experimental group, a 12-week/three-month physical activity coaching intervention will be conducted, while the control group will receive usual care. A post-intervention assessment will then be carried out, followed by follow-ups at 6 and 12 months after the baseline assessment.

The assessment will consist of a series of tests and questionnaires to record the following data: physical activity, functional capacity, muscle strength, health-related quality of life, symptoms, lung function, sociodemographic, and anthropometric data.

ELIGIBILITY:
Inclusion criteria:

* At least, 18 years of age.
* Having been diagnosed of COVID-19, confirmed by a polymerase chain reaction [PCR] test or an antigen test, at one of the severity levels during the acute phase of the illness.
* Presenting a diagnosis of post-COVID-19, persistent COVID, or long COVID, involving the persistence of symptoms for at least three months after the acute phase of the illness (i.e., to reduce variability in the diagnosis, it is proposed that symptom persistence be for at least 12 months).
* Being included in a post-COVID-19 follow-up consultation (or another consultation - pulmonology, internal medicine - in the event of closure of a specific consultation) in the region of Madrid, Spain.
* Stable condition of symptoms and comorbidities (i.e., no major change in clinical status).

Exclusion criteria:

* Presenting significant signs of cognitive decline, cardiovascular, neurological, and/or musculoskeletal disease that could hinder the performance of assessment tests and thus limit participation or pose a risk to their health.
* Particularly presenting the following conditions: cognitive disorders such as sequelae of Alzheimer's disease, senile dementia; comprehension disorders such as Wernicke's aphasia; cognitive-motor disorders such as hemiparesis/hemiplegia due to stroke; musculoskeletal disorders such as non-healed fractures, external prostheses (including prosthetic limbs for amputees); cardiovascular disorders such as unstable angina, recent acute myocardial infarction, among others.
* Medical history that interferes with the study's objectives or compromises its conclusions.
* Any health issues that limit life expectancy to less than one year.
* Medical, social, or geographical factor that may endanger the patient.
* Psycho-physical inability to complete assessment tests and questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Physical activity (PA) patterns (steps/day) from baseline (pre-intervention), at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Patients will wear an inertial measurement unit (a three-axial accelerometer and three-axial gyroscope) for one week. A valid assessment will require a minimum of four days with at least 8 hours of wearing time, excluding weekends.
  The minute-by-minute output, including the number of steps and metabolic equivalents of task (METs), will be exported.
  Using a statistical package and an appropriate algorithm, we will extract: the total daily step count (steps/day).
Change in Physical activity (PA) patterns (time spent in light PA per day) from baseline (pre-intervention), at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Patients will wear an inertial measurement unit (a three-axial accelerometer and three-axial gyroscope) for one week. A valid assessment will require a minimum of four days with at least 8 hours of wearing time, excluding weekends.
  The minute-by-minute output, including the number of steps and metabolic equivalents of task (METs), will be exported.
  Using a statistical package and an appropriate algorithm, we will extract: the total time spent in light PA per day (hours and minutes per day)
Change in Physical activity (PA) patterns (time spent in moderate-to-vigorous PA per day) from baseline (pre-intervention), at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Patients will wear an inertial measurement unit (a three-axial accelerometer and three-axial gyroscope) for one week. A valid assessment will require a minimum of four days with at least 8 hours of wearing time, excluding weekends.
  The minute-by-minute output, including the number of steps and metabolic equivalents of task (METs), will be exported.
  Using a statistical package and an appropriate algorithm, we will extract: the total time spent in moderate-to-vigorous PA per day (hours and minutes per day)
Change in Physical activity (PA) patterns (time in sedentary behaviour -lying or sitting- per day) from baseline (pre-intervention), at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Patients will wear an inertial measurement unit (a three-axial accelerometer and three-axial gyroscope) for one week. A valid assessment will require a minimum of four days with at least 8 hours of wearing time, excluding weekends.
  The minute-by-minute output, including the number of steps and metabolic equivalents of task (METs), will be exported.
  Using a statistical package and an appropriate algorithm, we will extract: the total time in sedentary behaviour -lying or sitting- per day (hours and minutes per day)
Change in functional capacity (six-minute walking test) from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Six-minute walking test/distance [6MWT/6MWD]. Patients will be asked to walk as far as possible in six minutes along a flat 30m corridor. Standardised instructions and encouragement will be given during the test, following European Respiratory Society/American Thoracic Society (ERS/ATS) statement.
Change in functional capacity (one-minute sit-to-stand test) from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  One-minute sit-to-stand [1minSTS]. Patients will sit and stand from a chair, without the aid of the upper limbs, many times as they can in a 1-min bout. Afterwards, the results will be compared to age- and sex-matched reference values.

SECONDARY OUTCOMES:
Change in isometric quadriceps strength from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Isometric quadriceps strength (dynamometer). A hand-held dynamometer will be used to assess isometric strength of the dominant leg. Participants will be seated at the edge of a treatment table, positioned at 60º of knee flexion, and with arms across the chest. The dynamometer will be positioned two fingers width above the lateral malleolus on the anterior aspect of the tibia.
  Four warm-ups will be allowed, on each at 25, 50, 75, and 100% of perceived effort, gradually building up to a maximal effort over 1 to 2 seconds.
  The tester will perform two make tests with the subject exerting 100% effort for 3 seconds. Average peak force of the two trials will be used to determine quadriceps muscle performance. The make test will entail the examiner giving appropriate resistance to the muscle force in order to ensure isometric conditions.
Change in handgrip force from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Handgrip force (dynamometer). A hand-held dynamometer will be used to measure isometric strength of the grip. Participants will be seated on a straight back chair with both feet flat on the floor. Arm positioning will be demonstrated by the examiner: the tested arm (dominant) will have the elbow bended to 90º, the forearm and wrist in neutral position, and the fingers flexed as needed for a maximal contraction, while the not-tested arm will assume an adducted and neutrally rotated shoulder position.
  Subjects will be instructed to breathe in through their nose and blow out through pursed lips while making a maximum grip effort. At this time, a verbal encouragement will be given by the examiner (e.g., "Squeeze! Harder! Harder! Relax!").
  Rest will be allowed between each grip assessment, no longer than four minutes. The average score among three trials will be recorded.
Change in maximal inspiratory and expiratory pressures from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Maximal respiratory pressures (PImax, PEmax) will be measured using a portable digital manometer; and assessed according to the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations [31] and following the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR) protocol.
  Then, the highest value of 3 attempts will be selected to obtain a reliable average, excluding pressure peaks lower than one second. Participants will be asked to sit with their neck and chest in an upright position and their feet flat on the floor. The results will be read using the current reference values in Spanish population provided by Lista-Paz et al. 2023.
Change in health-related quality of life from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Health-related quality of life [EuroQoL-five dimensions-five levels (EQ-5D-5L) questionnaire). The EQ-5D-5L consists of two parts: the descriptive system and a visual analogue scale (VAS). The descriptive system addresses five different dimensions (mobility, self-care, usual activities. pain/discomfort, and anxiety/depression), each with a five-point Likert-scale; the answering pattern can be transferred to a utility between 0 and 1 (the higher the better) by distinct (nation-specific) scoring algorithms. On the other hand, the VAS allows valuing current health on a 0-100 mm scale, with higher values indicating better health.
Change in dyspnoea symptom from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Dyspnea - modified Medical Research Council (mMRC) scale. The mMRC dyspnea scale consists of five grades of increasing severity. A higher score indicates a greater impact of dyspnea on activities of daily life.
Change in fatigue symptom from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Fatigue - Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale.
  The FACIT-F scale consists of many items to produce a global score, and each item can be scored from 0 to 4 (from "not at all" to "very much"). It covers different aspects of fatigue (physical, functional, emotional, and social consequences) with regard to the previous seven days. A higher score reflects less fatigue.
Change in anxiety and depression symptoms from baseline (pre-intervention) at 12 weeks (post-intervention), 6 months and 12 months | Baseline, 12 weeks, 6 months and 12 months
  Anxiety and depression-The Hospital Anxiety and Depression Scale (HADS). The HADS consists of two subscales (HADS-A, for anxiety disorders, and HADS-D, for depression) both containing seven intermingled items. A higher score implies a more severe case.
Forced expiratory volume in one second (FEV1) assessed using spirometry at baseline (pre-intervention). | Baseline.
  Forced expiratory volume in the first second (FEV1 in milliliters)
Forced expiratory volume in one second percentage predicted (FEV1%predicted) assessed using spirometry at baseline (pre-intervention). | Baseline.
  Forced expiratory volume in the first second (FEV1) as percentage predicted
Forced vital capacity (FVC) assessed using spirometry at baseline (pre-intervention). | Baseline.
  Forced vital capacity (FVC in milliliters)
Forced vital capacity percentage predicted (FVC%predicted) assessed using spirometry at baseline (pre-intervention). | Baseline.
  Forced vital capacity (FVC) as percentage predicted
Ratio between Forced expiratory volume in one second and Forced vital capacity (FEV1/FVC) assessed using spirometry at baseline (pre-intervention). | Baseline.
  Ratio between Forced expiratory volume in the first second and Forced vital capacity (FEV1/FVC, percentage)
Sociodemographics (age) at baseline (pre-intervention). | Baseline.
  Sociodemographics (age in years).
Sociodemographics (sex) at baseline (pre-intervention). | Baseline.
  Sociodemographics (sex, assessed as male/female).
Anthropometrics (height) at baseline (pre-intervention). | Baseline.
  Anthropometrics (height in meters).
Anthropometrics (weight) at baseline (pre-intervention). | Baseline.
  Anthropometrics (weight in kilograms).
Anthropometrics (body mass index - BMI) at baseline (pre-intervention). | Baseline.
  Weight and height will be combined to report BMI in kilograms/meters^2 (kg/m^2).
Proportion of participants with a diagnosed disease according to the International Classification of Diseases (ICD) at baseline (pre-intervention) | Baseline.
  Absolute and relative frequencies of any diagnosed disease will be reported using the International Classification of Diseases (ICD).
Proportion of participants following any pharmacological treatment or plan, as classified by the Anatomical Therapeutic Chemical (ATC) classification system at baseline (pre-intervention). | Baseline.
  Absolute and relative frequencies of any pharmacological treatment will be reported in accordance with the Anatomical Therapeutic Chemical (ATC) classification system.

CONTACTS AND LOCATIONS:
Overall Officials: María José Yuste Sánchez, PT, Ph.D., Principal Investigator — University of Alcalá, Alcalá de Henares (Madrid), Spain
Locations (1):
- University of Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after finalizing the draft of the database (at the end of follow-up), and only upon a formal request to the study principal investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available for one year after the final version of the database is considered complete.
Access Criteria: Formal request to the study principal investigator.

REFERENCES:
- [Background] Rabinovich RA, Louvaris Z, Raste Y, Langer D, Van Remoortel H, Giavedoni S, Burtin C, Regueiro EM, Vogiatzis I, Hopkinson NS, Polkey MI, Wilson FJ, Macnee W, Westerterp KR, Troosters T; PROactive Consortium. Validity of physical activity monitors during daily life in patients with COPD. Eur Respir J. 2013 Nov;42(5):1205-15. doi: 10.1183/09031936.00134312. Epub 2013 Feb 8. PMID 23397303
- [Background] Demeyer H, Burtin C, Van Remoortel H, Hornikx M, Langer D, Decramer M, Gosselink R, Janssens W, Troosters T. Standardizing the analysis of physical activity in patients with COPD following a pulmonary rehabilitation program. Chest. 2014 Aug;146(2):318-327. doi: 10.1378/chest.13-1968. PMID 24603844
- [Background] Taraldsen K, Chastin SF, Riphagen II, Vereijken B, Helbostad JL. Physical activity monitoring by use of accelerometer-based body-worn sensors in older adults: a systematic literature review of current knowledge and applications. Maturitas. 2012 Jan;71(1):13-9. doi: 10.1016/j.maturitas.2011.11.003. Epub 2011 Nov 30. PMID 22134002
- [Background] Demeyer H, Burtin C, Hornikx M, Camillo CA, Van Remoortel H, Langer D, Janssens W, Troosters T. The Minimal Important Difference in Physical Activity in Patients with COPD. PLoS One. 2016 Apr 28;11(4):e0154587. doi: 10.1371/journal.pone.0154587. eCollection 2016. PMID 27124297
- [Background] Gardner AW, Montgomery PS, Wang M, Shen B. Minimal clinically important differences in daily physical activity outcomes following supervised and home-based exercise in peripheral artery disease. Vasc Med. 2022 Apr;27(2):142-149. doi: 10.1177/1358863X211072913. Epub 2022 Feb 15. PMID 35164605
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. doi: 10.2466/pms.1995.80.1.163. PMID 7624188
- [Background] Vaidya T, de Bisschop C, Beaumont M, Ouksel H, Jean V, Dessables F, Chambellan A. Is the 1-minute sit-to-stand test a good tool for the evaluation of the impact of pulmonary rehabilitation? Determination of the minimal important difference in COPD. Int J Chron Obstruct Pulmon Dis. 2016 Oct 19;11:2609-2616. doi: 10.2147/COPD.S115439. eCollection 2016. PMID 27799759
- [Background] Deones VL, Wiley SC, Worrell T. Assessment of quadriceps muscle performance by a hand-held dynamometer and an isokinetic dynamometer. J Orthop Sports Phys Ther. 1994 Dec;20(6):296-301. doi: 10.2519/jospt.1994.20.6.296. PMID 7849749
- [Background] Oliveira A, Rebelo P, Paixao C, Jacome C, Cruz J, Martins V, Simao P, Brooks D, Marques A. Minimal Clinically Important Difference for Quadriceps Muscle Strength in People with COPD following Pulmonary Rehabilitation. COPD. 2021 Feb;18(1):35-44. doi: 10.1080/15412555.2021.1874897. Epub 2021 Feb 3. PMID 33533285
- [Background] Hamilton GF, McDonald C, Chenier TC. Measurement of grip strength: validity and reliability of the sphygmomanometer and jamar grip dynamometer. J Orthop Sports Phys Ther. 1992;16(5):215-9. doi: 10.2519/jospt.1992.16.5.215. PMID 18796752
- [Background] Bohannon RW. Minimal clinically important difference for grip strength: a systematic review. J Phys Ther Sci. 2019 Jan;31(1):75-78. doi: 10.1589/jpts.31.75. Epub 2019 Jan 10. PMID 30774209
- [Background] Lista-Paz A, Langer D, Barral-Fernandez M, Quintela-Del-Rio A, Gimeno-Santos E, Arbillaga-Etxarri A, Torres-Castro R, Vilaro Casamitjana J, Varas de la Fuente AB, Serrano Veguillas C, Bravo Cortes P, Martin Cortijo C, Garcia Delgado E, Herrero-Cortina B, Valera JL, Fregonezi GAF, Gonzalez Montanez C, Martin-Valero R, Francin-Gallego M, Sanesteban Hermida Y, Gimenez Moolhuyzen E, Alvarez Rivas J, Rios-Cortes AT, Souto-Camba S, Gonzalez-Doniz L. Maximal Respiratory Pressure Reference Equations in Healthy Adults and Cut-off Points for Defining Respiratory Muscle Weakness. Arch Bronconeumol. 2023 Dec;59(12):813-820. doi: 10.1016/j.arbres.2023.08.016. Epub 2023 Sep 29. English, Spanish. PMID 37839949
- [Background] Szentes BL, Kreuter M, Bahmer T, Birring SS, Claussen M, Waelscher J, Leidl R, Schwarzkopf L. Quality of life assessment in interstitial lung diseases:a comparison of the disease-specific K-BILD with the generic EQ-5D-5L. Respir Res. 2018 May 25;19(1):101. doi: 10.1186/s12931-018-0808-x. PMID 29801506
- [Background] Garcia-Gordillo MA, Adsuar JC, Olivares PR. Normative values of EQ-5D-5L: in a Spanish representative population sample from Spanish Health Survey, 2011. Qual Life Res. 2016 May;25(5):1313-21. doi: 10.1007/s11136-015-1164-7. Epub 2015 Oct 19. PMID 26482825
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Hewlett S, Dures E, Almeida C. Measures of fatigue: Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire (BRAF MDQ), Bristol Rheumatoid Arthritis Fatigue Numerical Rating Scales (BRAF NRS) for severity, effect, and coping, Chalder Fatigue Questionnaire (CFQ), Checklist Individual Strength (CIS20R and CIS8R), Fatigue Severity Scale (FSS), Functional Assessment Chronic Illness Therapy (Fatigue) (FACIT-F), Multi-Dimensional Assessment of Fatigue (MAF), Multi-Dimensional Fatigue Inventory (MFI), Pediatric Quality Of Life (PedsQL) Multi-Dimensional Fatigue Scale, Profile of Fatigue (ProF), Short Form 36 Vitality Subscale (SF-36 VT), and Visual Analog Scales (VAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S263-86. doi: 10.1002/acr.20579. No abstract available. PMID 22588750
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Smid DE, Franssen FM, Houben-Wilke S, Vanfleteren LE, Janssen DJ, Wouters EF, Spruit MA. Responsiveness and MCID Estimates for CAT, CCQ, and HADS in Patients With COPD Undergoing Pulmonary Rehabilitation: A Prospective Analysis. J Am Med Dir Assoc. 2017 Jan;18(1):53-58. doi: 10.1016/j.jamda.2016.08.002. Epub 2016 Sep 10. PMID 27624705